CLINICAL TRIAL: NCT03537053
Title: Exploring the Acceptability of "Move a Little and Often"- a Behaviour Change Intervention to Reduce Sedentary Behaviours in People With Long Term Conditions and Symptoms of Depression.
Brief Title: An Approach to "Move a Little & Often" With Health Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Isabel Adeyemi, Principle Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS ID: 244602
Record Dates: First submitted 2018-05-01; First posted 2018-05-25 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Depression; Multiple Chronic Conditions
Keywords: Sedentary Lifestyle
MeSH Terms: conditions — Depression; Multiple Chronic Conditions; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: a single group feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A plan to Move a Little and Often (Experimental): The intervention will consist of 3 components: a short video will raise awareness about the impact of sedentary behaviours, a booklet, and an online forum on Facebook to encourage participants to support each other.
  At the end of the baseline data collection, participants will be asked to watch the video. They will then be given the booklet and invited to join the Facebook group. A minimum of 5 participants must be recruited prior to running the Facebook group.
  Interventions: Behavioral: A plan to Move a Little and Often

INTERVENTIONS:
Behavioral: A plan to Move a Little and Often — The intervention content is reported using the behaviour change technique (BCT) Taxonomy v1 (Michie, et al. 2013). The video will contain the BCT: information about health consequences. The booklet will consist of BCTs: self-monitoring of behaviour, goal setting behaviour, action planning, commitment, social support (practical), self-talk, and mental rehearsal of successful performance. Lastly, usage of the Facebook group will include BCTs: commitment, and social support unspecified, practical and emotional.
  Mental rehearsal, goal setting behaviour and action planning will be delivered through mental simulation exercises (Taylor, et al. 1998). BCTs self-monitoring of behaviour, goal setting behaviour, and commitment will be delivered using implementation intentions (Gollwitzer 1993).

SUMMARY:
People with long term conditions such as diabetes and arthritis, and who also have depression spend a lot of time sedentary during the day. This is because they face many barriers to being active, such as pain and fatigue. Being sedentary is problematic because it is associated with poorer health in the long term.

Common sedentary behaviours are watching television and using the computer; these behaviours are labelled as screen-based sedentary behaviours. An intervention to reduce these behaviours could improve mental and physical wellbeing. The aim of the study is to explore the acceptability of an intervention to "Move a Little and Often" in people with depression symptoms and long term conditions. The investigators will explore the intervention's acceptability using interviews and will examine if the intervention is associated with a reduction in time spent sedentary. Results will help refine the intervention further.

The feasibility study is part of a PhD project funded by the National Institute of Health Research (NIHR) Collaborations for Leadership in Applied Health Research and Care (CLAHRC) Greater Manchester

DETAILED DESCRIPTION:
There is a growing focus in research on the need to reduce sedentary behaviours. Studies have shown that independently of moderate to vigorous physical activity, the amount of time spent sedentary predicts poorer health outcomes. This means that in addition to exercising, it is important to reduce prolonged periods of sedentary behaviours to improve health. For people with depression and long term conditions, milder forms of physical activity may be more appropriate due to higher levels of pain and fatigue resulting from exercise. Reducing sedentary behaviours by substituting them with mild physical activities such as walking is a potential avenue to improve health outcomes in this population group.

To date, no intervention has been developed to reduce prolonged periods of sedentariness in people with depression and long term health conditions within the UK. This feasibility study aims to refine a behaviour change intervention to reduce sedentary time in this population group. The intervention has been developed through reviewing the literature on interventions to increase physical activity (a systematic review), an interview study to explore sedentary and physical activity behaviours within this population group, and through patient and public involvement.

ELIGIBILITY:
Inclusion Criteria:

* be aged ≥18 years,
* self-report a clinical diagnosis of a long term physical health condition;
* score 8 or more on the depression subscale of the Hospital hospital anxiety and depression scales (Zigmond & Snaith, 1983) suggesting the presence of depression;
* speak English fluently;
* live within Greater Manchester

Exclusion Criteria:

* are not registered with a GP practice,
* in receipt of palliative care,
* report a diagnosis of severe mental health problems such as schizophrenia or bipolar disorder,
* have had a recent bereavement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
The short form International Physical Activity Questionnaire (IPAQ ; Booth 2000). | 1 month follow-up
  The IPAQ will be used to measure frequency and duration of sedentariness, and any increase in physical activity. The IPAQ asks about walking, moderate intensity activities and vigorous-intensity activities. In order to compute the total score, it requires summation of the durations (minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.

OTHER OUTCOMES:
Sedentary Behaviour Questionnaire (Gardiner, et al. 2011) | 1 month follow-up
  The Sedentary Behaviour Questionnaire is a seven-item questionnaire that asks participants to report on activities they did during the last week while they were sitting or lying down, and to report the total time spent in each activity. The seven individual sedentary items are TV or video/DVD watching, computer use, reading, socializing with friends or family, time traveling in a motor vehicle or on public transport, doing hobbies, and any other activities they did while they were sitting or lying down. The measure has previously been used in a study of sedentariness in older adults (Gardiner, et al. 2011).
The International Sedentary Assessment Tool (ISAT; Prince, et al. 2017) | 1 month follow-up
  The ISAT contains 5 items relating to total time spent sedentary and time spent doing specific activities: television use, computer use, using transport, and reading. Participants will be asked how much time they spend on each activity over the course of a typical week. Psychometric properties have yet to be reported for this questionnaire measure.
The Hospital Anxiety and Depression Scale (HADS; Zigmond and Snaith 1983) | 1 month follow-up
  The HADS will measure depression and anxiety. The HADS is a 14-item self-report screening scale for anxiety and depression symptoms. It contains two 7 item scales: one for anxiety and one for depression; both of which have a score ranging from 0-21. The HADS is commonly used in research studies and has good validity (Bjelland et al. 2002, et al. 2005).
The Numeric Rating Scale (NRS; Herr and Mobily 1993). | 1 month follow-up
  Pain will be measured using the 0-10 Numeric Rating Scale (NRS) (Herr and Mobily 1993). Participants will be asked to rate their pain over the previous week. This questionnaire has been found to correlate significantly with other pain measures (Herr, et al. 2004). Scores can range from 0 to 10, with higher scores indicating more pain.
The Pittsburgh Sleep Quality Index (Buysse, et al. 1989) | 1 month follow-up
  Sleep quality and disturbances will be measured using the Pittsburgh Sleep Quality Index (Buysse, et al. 1989). The questionnaire can be used to generate seven component scores for subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each of the seven component scores is weighted equally on a scale of 0 (no difficulty) to 3 (severe difficulty). The seven component scores are then summed to yield a global PSQI score, ranging from 0 to 21, with a higher score indicating poorer sleep quality.
The Measure of National Wellbeing (Carter 2017) | 1 month follow-up
  Quality of life will be measured using items from the Measure of National Wellbeing used by the Office for National Statistics. Participants will be asked: overall, how satisfied they are with life nowadays; overall, to what extent they feel the things they do in life are worthwhile; overall, how happy they felt yesterday; overall, how anxious they felt yesterday?. Each question is answered on a scale of 0 to 10. People are asked to respond on a scale of 0 to 10, where 0 is "not at all" and 10 is "completely". Mean ratings for all 4 personal well-being questions will be calculated.
Short Form Health Survey (SF-12; Ware, et al. 1996) | 1 month follow-up
  The SF 12 is a 12 item measure with two scales: mental and physical functioning and overall health-related-quality of life. The SF-12 is weighted and summed to provide Physical and Mental Health Composite Scores (PCS & MCS). These two composite scores are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The questionnaire was adapted from the SF-36 Health Survey and its results can be compared with the SF36 (Jenkinson, et al. 1997)
The ENRICHD Social Support Instrument (Mitchell, et al. 2003) | 1 month follow-up
  Social support will be measured using the ENRICHD Social Support Instrument (Mitchell, et al. 2003). The ENRICHD Social Support Instrument (ESSI) is a brief seven-item measure of perceived social support. The scale contains six social support items that have been shown to be individually predictive of poor outcome in patients with cardiac disease, and one item that assesses partner status.
The Self-Report Behavioural Automaticity Index SRBAI (Gardner, et al. 2012) | 1 month follow-up
  The SRBAI will be used to measure habit strength for avoiding sedentariness. Participants will be asked to rate 4 items on a Likert scale of 0 (strongly disagree) to 5 (strongly agree). The 4 items are: avoiding being sedentary is something:- 1) I do automatically; 2) I do without having to consciously remember,3) I do without thinking, 4) I start doing before I realise I'm doing it.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Adeyemi, MPhil, Principal Investigator — The University of Manchester
Locations (2):
- United Kingdom (2):
  - The University of Manchester, Manchester
  - Salford Royal NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data on demographics (age, gender) and standardised questionnaire measures will be shared.
Supporting Information: Study Protocol
Time Frame: The data will become available upon publication of the study in an academic journal.